CLINICAL TRIAL: NCT00729443
Title: A Single-Centre, Placebo-Controlled, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD3241 Following Administration of Single Ascending (Part A) and Fractionated Ascending (Part B) Oral Doses to Young Healthy Volunteers
Brief Title: Investigating Safety, Tolerability and Pharmakinetics When Giving Single and Fractionated Doses of AZD3241 to Healthy Volunteers
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jarkko Kalliomäki, MD, Medical Science Director, Neuroscience alpha, AstraZeneca R&D Södertälje, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0490C00012; EudractCT# 2008-002466-62
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Volunteers
Keywords: Single dose; Phase 1; Safety of AZD3241; tolerability of AZD3241
MeSH Terms: interventions — AZD3241

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD3241
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3241 — single oral dose
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The study is carried out in order to investigate safety, tolerability and pharmacokinetics after administrating single and fractionated doses of AZD3241 to healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Body Mass Index (BMI) 19 to 30 kg/m2 inclusive
* Clinically normal physical findings, including BP, pulse rate, ECG and laboratory findings, as judged by the investigator

Exclusion Criteria:

* Clinically significant illness within the 2 weeks prior to the administration of the investigational product
* Heart rate (resting, recumbent) <50 bmp or >85 bmp
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity as judged by the investigator

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
General tolerability and safety variables | 2 weeks

SECONDARY OUTCOMES:
pk | approximately 48 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Bylesjö, Principal Investigator — Astrazeneca Clinical Pharmacology Unit, Stockholm, Sweden
Locations (1):
- Research Site, Stockholm, Sweden